CLINICAL TRIAL: NCT05446857
Title: Glecaprevir/Pibrentasvir for the Treatment of PTSD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bradley Watts, Staff Psychiatrist, White River Junction Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1673711
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: PTSD
Keywords: PTSD; Antiviral; Hepatitis C
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Hepatitis C | interventions — glecaprevir; pibrentasvir; glecaprevir and pibrentasvir

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Active Drug (Experimental): All enrolled participants will receive Glecaprevir/Pibrentasvir
  Interventions: Drug: Glecaprevir / Pibrentasvir Pill

INTERVENTIONS:
Drug: Glecaprevir / Pibrentasvir Pill — Glecaprevir 100 mg/Pibrentasvir 40 mg, 3 oral tablets once daily for 8 weeks.
  Other Names: Mavyret

SUMMARY:
An open-label pilot study to further investigate glecaprevir/pibrentasvir (GLE/PIB), a direct acting antiviral (DAA) that has been associated with posttraumatic stress disorder (PTSD) symptom improvement when prescribed for the treatment of chronic hepatitis C viral infection (HCV).

DETAILED DESCRIPTION:
To perform an open-label pilot study (N=10) to further investigate glecaprevir/pibrentasvir (GLE/PIB), a direct acting antiviral (DAA) that has been associated with posttraumatic stress disorder (PTSD) symptom improvement when prescribed for the treatment of chronic hepatitis C viral infection (HCV). The specific research described in this proposal is intended to pilot GLE/PIB for N=10 patients with PTSD in the absence of HCV.

Primary Aims:

Aim 1: Determine the feasibility of testing GLE/PIB for PTSD symptoms. Aim 2: Determine the feasibility of testing GLE/PIB for functioning among patients with PTSD.

Aim 3: Assess the safety and tolerability of GLE/PIB treatment for patients with PTSD in the absence of HCV.

Exploratory Aim: Investigate the possible biological mechanism of GLE/PIB for PTSD via blood bio-marker analyses.

ELIGIBILITY:
Inclusion Criteria Summary

1. Age 19-70 years
2. Weight ≥ 45 kg
3. PTSD as determined by the CAPS within seven days of enrollment.
4. Eligible for Veterans Affairs healthcare.
5. If of childbearing potential, use of acceptable method of birth control (i.e., effective contraceptives, abstinence) is required.
6. Able to read, understand, and sign the informed consent document.

Exclusion Criteria:

1. Pregnant or lactating person
2. Moderate or severe hepatic impairment (Child-Pugh B or C)
3. History of prior hepatic decompensation
4. Current use of drugs listed as having significant drug interactions on prescribing label
5. Advanced liver disease
6. Current or prior hepatitis B infection
7. Prior clinical use of GLE/PIB or HCV NS5A inhibitor AND NS3/4A protease inhibitor
8. Current HCV infection
9. Current psychosis or mania
10. Significant suicidal ideation
11. Unstable medical conditions
12. Current severe alcohol or substance use disorder (excluding nicotine)
13. Evidence-based PTSD psychotherapy changes in the past two months
14. Evidence-based PTSD medication changes in the past two months

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Clinical Administered Post-Traumatic Stress Disorder Scale version 5 (CAPS-5) | Change from Baseline CAPS score at 8 weeks
  Queries the frequency and intensity of symptoms of Post-traumatic Stress Disorder (PTSD). The score ranges from 0-80 with a higher score indicating worse symptoms. It is considered the gold standard for diagnosis and symptoms assessment in PTSD clinical studies.
World Health Organization Disability Assessment Schedule, version 2.0 (WHODAS) | Change from Baseline WHODAS score at 8 weeks
  A 36 item self-report instrument that assesses disability and function across six domains: communicating, getting around, self-care, getting along with people, life activities, and participation in society. The WHODAS has been used as an outcome of function and disability across many disorders and is commonly used in mental health treatment trials. The total score ranges from 0-180 with a higher score indicating worse functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley V Watts, MD, MPH, Principal Investigator — White River Junction Veterans Affairs Medical Center
Locations (1):
- White River Junction VAMC, White River Junction, Vermont, United States

IPD SHARING:
Plan to Share IPD: No